CLINICAL TRIAL: NCT02710045
Title: The Interaction Between Live and Killed Vaccines: the Effect of the Diphtheria-tetanus-whole Cell Pertussis (DTP) Combined Vaccine on T Cell Memory Following Measles Vaccination
Brief Title: The Interaction Between Measles and DTP Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Unit, The Gambia (Other)
Responsible Party: Sponsor
Organization: London School of Hygiene and Tropical Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SCC 1085
Record Dates: First submitted 2016-03-03; First posted 2016-03-16 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-12

CONDITIONS: Non-target Heterologous Effects of Vaccines; Vaccine Interactions
Keywords: Immunity, Innate; Immunity, Non-Specific; Antibodies; Cytokines; Immunity, Cellular
MeSH Terms: interventions — Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MV at 9 months (Active Comparator): Measles Vaccine at 9 months of age. Measles Vaccine at 18 months of age. All vaccines given as per normal Gambia schedule until 9 months of age, including third dose of diphtheria-tetanus-whole cell pertussis (DTP3), hepatitis B vaccine (HBV) and oral polio vaccine (OPV) at four months of age.
  At 9 months of age given a single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid. Yellow fever vaccine (YF) and OPV administered at 11 months of age. Given a standard MV challenge at 18 months of age.
  Interventions: Biological: Measles Vaccine at 9 months of age; Biological: Measles Vaccine at 18 months of age
- DTP + MV at 9 months (Active Comparator): Measles Vaccine at 9 months of age. DTP Vaccine at 9 months of age. Measles Vaccine at 18 months of age. DTP3 dose withheld and given HBV and OPV at four months of age. At 9 months of age given a single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid, and i.m. DTP (Serum Institute of India Ltd.) in the thigh. Yellow fever vaccine (YF) and OPV administered at 11 months of age. Given a standard MV challenge at 18 months of age.
  Interventions: Biological: Measles Vaccine at 9 months of age; Biological: DTP Vaccine at 9 months of age; Biological: Measles Vaccine at 18 months of age
- DTP at 9 months (Active Comparator): DTP Vaccine at 9 months of age. Measles Vaccine at 18 months of age. DTP3 dose withheld and given HBV and OPV at four months of age. At 9 months of age given i.m. DTP (Serum Institute of India Ltd.) in the thigh. MV, OPV and YF administered at 11 months of age. Given a standard MV challenge at 18 months of age.
  Interventions: Biological: DTP Vaccine at 9 months of age; Biological: Measles Vaccine at 18 months of age

INTERVENTIONS:
Biological: Measles Vaccine at 9 months of age — Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 9 months of age
  Other Names: MV
  Arms: DTP + MV at 9 months; MV at 9 months
Biological: DTP Vaccine at 9 months of age — Single intramuscular (i.m.) dose of diphtheria-tetanus-whole cell pertussis vaccine (Serum Institute of India Ltd.) into the thigh at 9 months of age
  Other Names: DTP
  Arms: DTP + MV at 9 months; DTP at 9 months
Biological: Measles Vaccine at 18 months of age — Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 18 months of age
  Other Names: MV

SUMMARY:
The purpose of this study is to investigate for the broad immunological effects of administering measles vaccine (MV) and diphtheria-tetanus-whole cell pertussis vaccine (DTP) to 9 month old Gambian infants, either alone or together. Effects on vaccine-specific immune responses, innate immunity, and immune memory were studied. The hypothesis is that when MV and DTP are given together there will be more inflammation and this will interfere with generation of immunity to the vaccine and to other non-vaccine related stimuli.

DETAILED DESCRIPTION:
Many studies demonstrate that routine Expanded Program on Immunisation (EPI) vaccinations have "non-specific" or "heterologous" effects on child survival that cannot be accounted for by protection against the vaccine specific disease. These effects were overlooked in the past because it was assumed that the impact on survival would be proportional to reduction in the targeted infection. Large epidemiological studies in Bangladesh and Guinea-Bissau have shown that live vaccines, including measles vaccine (MV), have beneficial effects on overall mortality which cannot be explained by protection against the vaccine specific disease. Deleterious non-specific effects were shown convincingly in the high-titre MV trials in which girls, but not boys, had a two-fold increase in mortality even though the vaccine was fully protective against measles. A reinterpretation of these trials indicated that the most likely explanation was that the increased female mortality was due to inactivated vaccines provided after MV. It has further been shown in smaller observational studies that receiving diphtheria, tetanus and whole cell pertussis combined vaccine (DTwP) either with or after MV negates the beneficial effects of MV, and may lead to increased mortality. However, the increased mortality of girls in male-female twin pairs was not apparent when MV was given after the last dose of DTwP. In the present EPI schedule in The Gambia, DTwP is administered as a single dose vaccine at 2, 3 and 4 months, and MV at nine months. However, many children, particularly in low income countries, present late for their vaccines and may subsequently receive them in the wrong order. In particular DTP is often given at the wrong time point, e.g. the third DTP dose (DTP3) with MV. Given the increasing evidence that the order in which vaccines are administered is crucial, the routine practice of administering missed EPI vaccines at late presentation or boosting with DTP in year 2 may not be advisable.

The mechanism behind these effects is unknown, and whether there is an immunological basis has yet to be explored. The majority of controlled trials of vaccine efficacy have focused on vaccine specific antibody (Ab) responses to test vaccine efficacy, and few studies have investigated T cell memory induction, despite the fact that it is likely to be critical for long term protection. Indeed, the cellular response to MV seems to be crucial in protecting against severe disease and death, and cellular responses are required to protect against Bordetella pertussis infection. Live vaccines such as bacillus Calmette-Guerin (BCG) and MV have been shown to stimulate Th1 type immune responses. The immune response to DTwP, a killed vaccine, tends to be Th2 biased in early life, despite the fact that the whole cell pertussis component biases towards a Th1 response. DTwP contains an aluminium based adjuvant, aluminium hydroxide, which is excellent at promoting humoral and Th2 responses, but poor at generating good cell mediated immunity and long term T cell memory. This polarisation of cellular reactivity to live and killed vaccines may explain why administering a killed vaccine with a live vaccine abrogates the beneficial effect of the live vaccine. Conversely, administering a live vaccine after DTwP may cause a shift towards protective Th1 type immunity, thus diminishing the harmful effects of DTwP and providing a non-specific survival benefit. Interestingly, aluminium hydroxide has been shown to cause enhanced susceptibility to tuberculosis (TB) in animal models. Thus the aluminium adjuvant in DTwP may play a role in the deleterious effect of DTwP on live vaccines, possibly through an influence on the generation of T cell memory to other infections and vaccines.

Attributing the observed effects of the DTwP / MV interactions entirely to shifts in the T helper cell 1 (Th1) / Th2 profile is likely to be an over simplification, but provides a good starting point for unravelling this phenomenon. Other arms of the immune response that need to be considered are regulatory T cells (Tregs) and the Th17 inflammatory T cell lineage. The former are a heterogeneous group of naturally occurring and induced T cells, and have been shown to play a regulatory role in immunity to a number of infectious diseases, but almost nothing is known about their generation or functional role in vaccine immunogenicity in humans. Newborns are known to have high levels of functional Tregs, and these are likely to be essential in controlling the immune response to antigens encountered in early life, as well as modulating self reactive responses. Measles vaccination causes suppression of T cell responses, and measles vaccinated children upregulate Forkhead Box P3 (FOXP3) expression (Ota et al, personal communication), suggesting a role for Tregs. Thus Treg induction is likely to be an important component of the immune response to MV.

This study will investigate in detail the immunological consequences of giving DTP or MV alone or at the same time. The study will involve an intervention trial to analyse the effect of giving DTP with MV on the generation of T cell memory (effector and central), humoral responses, pro-inflammatory cytokine profile (Th1, Th2, Th17) and Treg responses to measles and recall antigens. Our detailed immunological studies will provide vital immunological data on potential mechanisms of the DTP / MV interaction. A comprehensive understanding of the immunological effects of administering either DTP alone or DTP and MV simultaneously will help us understand why these interventions might be detrimental, and may suggest the need to refine current EPI practices. It is also crucial to gain a detailed understanding of the immunological effects of possible deleterious interactions between the current EPI vaccines, before introducing new vaccines that are becoming available for testing in early life e.g. TB and malaria vaccines. Furthermore, understanding mechanisms whereby MV provides survival benefits might identify strategies that can be harnessed in future vaccine design.

All infants will be given a MV challenge at 18 months of age and immunological parameters will be analysed 1 month later. This will establish whether any vaccine group effects at 10 months off age persist until 18 months of age and influence the immune response to a new immune challenge.

Two primary hypotheses as detailed below will be tested as a starting point, but other immunological assays will be conducted. Furthermore all analyses will take sex into account since the heterologous effects of vaccines are different in males and females, with females generally being more susceptible.

Hypotheses:

1. DTP (a killed vaccine) drives primarily a Th2 response and MV (a live vaccine) drives primarily a Th1 response. A DTP driven Th2 response occurring at the time of trying to activate a Th1 response to MV will interfere with the priming of measles specific memory responses and responses to other recall antigens.
2. The extra Th2 stimulation from DTP at the time of MV will provide too many signals to allow the generation of regulatory T cells (Tregs) which are an essential component of the immunological response to MV.

ELIGIBILITY:
* Inclusion Criteria:

  * Healthy 4 month old infants
  * All EPI vaccines received to date according to current Gambia government schedule
  * Normal weight for age according to growth chart
* Exclusion Criteria:

  * Temperature >37.5°C
  * Any history of ongoing chronic illness

Ages: 16 Weeks to 22 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie L Flanagan, PhD, Principal Investigator — University of Tasmania, Australia

IPD SHARING:
Plan to Share IPD: No
The data will be made available upon written request

REFERENCES:
- [Background] Aaby P, Jensen H, Samb B, Cisse B, Sodemann M, Jakobsen M, Poulsen A, Rodrigues A, Lisse IM, Simondon F, Whittle H. Differences in female-male mortality after high-titre measles vaccine and association with subsequent vaccination with diphtheria-tetanus-pertussis and inactivated poliovirus: reanalysis of West African studies. Lancet. 2003 Jun 28;361(9376):2183-8. doi: 10.1016/S0140-6736(03)13771-3. PMID 12842371
- [Background] Kristensen I, Aaby P, Jensen H. Routine vaccinations and child survival: follow up study in Guinea-Bissau, West Africa. BMJ. 2000 Dec 9;321(7274):1435-8. doi: 10.1136/bmj.321.7274.1435. PMID 11110734
- [Background] Aaby P, Jensen H, Gomes J, Fernandes M, Lisse IM. The introduction of diphtheria-tetanus-pertussis vaccine and child mortality in rural Guinea-Bissau: an observational study. Int J Epidemiol. 2004 Apr;33(2):374-80. doi: 10.1093/ije/dyh005. PMID 15082643
- [Background] Veirum JE, Sodemann M, Biai S, Jakobsen M, Garly ML, Hedegaard K, Jensen H, Aaby P. Routine vaccinations associated with divergent effects on female and male mortality at the paediatric ward in Bissau, Guinea-Bissau. Vaccine. 2005 Jan 19;23(9):1197-204. doi: 10.1016/j.vaccine.2004.02.053. PMID 15629363
- [Background] Permar SR, Klumpp SA, Mansfield KG, Carville AA, Gorgone DA, Lifton MA, Schmitz JE, Reimann KA, Polack FP, Griffin DE, Letvin NL. Limited contribution of humoral immunity to the clearance of measles viremia in rhesus monkeys. J Infect Dis. 2004 Sep 1;190(5):998-1005. doi: 10.1086/422846. Epub 2004 Jul 26. PMID 15295708
- [Background] Mills KH, Ryan M, Ryan E, Mahon BP. A murine model in which protection correlates with pertussis vaccine efficacy in children reveals complementary roles for humoral and cell-mediated immunity in protection against Bordetella pertussis. Infect Immun. 1998 Feb;66(2):594-602. doi: 10.1128/IAI.66.2.594-602.1998. PMID 9453614
- [Background] Ovsyannikova IG, Reid KC, Jacobson RM, Oberg AL, Klee GG, Poland GA. Cytokine production patterns and antibody response to measles vaccine. Vaccine. 2003 Sep 8;21(25-26):3946-53. doi: 10.1016/s0264-410x(03)00272-x. PMID 12922130
- [Background] Rowe J, Macaubas C, Monger T, Holt BJ, Harvey J, Poolman JT, Loh R, Sly PD, Holt PG. Heterogeneity in diphtheria-tetanus-acellular pertussis vaccine-specific cellular immunity during infancy: relationship to variations in the kinetics of postnatal maturation of systemic th1 function. J Infect Dis. 2001 Jul 1;184(1):80-8. doi: 10.1086/320996. Epub 2001 May 29. PMID 11398113
- [Background] Lavigne MV, Castro M, Mateo N, Deluchi S, Atzori C, Piudo L, Calcagno M, Brero ML, Manghi M. Whole-cell Bordetella pertussis vaccine component modulates the mouse immune response to an unrelated soluble antigen. Microbes Infect. 2002 Jul;4(8):815-20. doi: 10.1016/s1286-4579(02)01601-5. PMID 12270728
- [Background] Lindblad EB. Aluminium compounds for use in vaccines. Immunol Cell Biol. 2004 Oct;82(5):497-505. doi: 10.1111/j.0818-9641.2004.01286.x. PMID 15479435
- [Background] Lindblad EB, Elhay MJ, Silva R, Appelberg R, Andersen P. Adjuvant modulation of immune responses to tuberculosis subunit vaccines. Infect Immun. 1997 Feb;65(2):623-9. doi: 10.1128/iai.65.2.623-629.1997. PMID 9009322
- [Background] Weaver CT, Harrington LE, Mangan PR, Gavrieli M, Murphy KM. Th17: an effector CD4 T cell lineage with regulatory T cell ties. Immunity. 2006 Jun;24(6):677-688. doi: 10.1016/j.immuni.2006.06.002. PMID 16782025
- [Background] Baecher-Allan C, Viglietta V, Hafler DA. Human CD4+CD25+ regulatory T cells. Semin Immunol. 2004 Apr;16(2):89-98. doi: 10.1016/j.smim.2003.12.005. PMID 15036232
- [Background] Mills KH. Regulatory T cells: friend or foe in immunity to infection? Nat Rev Immunol. 2004 Nov;4(11):841-55. doi: 10.1038/nri1485. PMID 15516964
- [Background] Smedman L, Joki A, da Silva AP, Troye-Blomberg M, Aronsson B, Perlmann P. Immunosuppression after measles vaccination. Acta Paediatr. 1994 Feb;83(2):164-8. doi: 10.1111/j.1651-2227.1994.tb13043.x. PMID 8193495
- [Background] Pala S, Crimaldi G, Consolini R, Macchia P. [The cell-mediated response after measles vaccination]. Pediatr Med Chir. 1998 May-Jun;20(3):213-6. Italian. PMID 9744016
- [Background] Sallusto F, Geginat J, Lanzavecchia A. Central memory and effector memory T cell subsets: function, generation, and maintenance. Annu Rev Immunol. 2004;22:745-63. doi: 10.1146/annurev.immunol.22.012703.104702. PMID 15032595
- [Background] Aaby P, Bhuiya A, Nahar L, Knudsen K, de Francisco A, Strong M. The survival benefit of measles immunization may not be explained entirely by the prevention of measles disease: a community study from rural Bangladesh. Int J Epidemiol. 2003 Feb;32(1):106-16. doi: 10.1093/ije/dyg005. PMID 12690020
- [Background] Aaby MP, Samb B, Simondon F, Seck AM, Knudsen KM, Whittle H. [A non-specific, beneficial effect of measles vaccination. Analysis of mortality studies from developing countries]. Ugeskr Laeger. 1996 Oct 14;158(42):5944-8. Danish. PMID 8928283
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Pulendran B. Systems vaccinology: probing humanity's diverse immune systems with vaccines. Proc Natl Acad Sci U S A. 2014 Aug 26;111(34):12300-6. doi: 10.1073/pnas.1400476111. Epub 2014 Aug 18. PMID 25136102
- [Background] Li S, Nakaya HI, Kazmin DA, Oh JZ, Pulendran B. Systems biological approaches to measure and understand vaccine immunity in humans. Semin Immunol. 2013 Oct 31;25(3):209-18. doi: 10.1016/j.smim.2013.05.003. Epub 2013 Jun 21. PMID 23796714
- [Background] Flanagan KL, Klein SL, Skakkebaek NE, Marriott I, Marchant A, Selin L, Fish EN, Prentice AM, Whittle H, Benn CS, Aaby P. Sex differences in the vaccine-specific and non-targeted effects of vaccines. Vaccine. 2011 Mar 16;29(13):2349-54. doi: 10.1016/j.vaccine.2011.01.071. Epub 2011 Feb 5. PMID 21300095
- [Background] Klein SL, Jedlicka A, Pekosz A. The Xs and Y of immune responses to viral vaccines. Lancet Infect Dis. 2010 May;10(5):338-49. doi: 10.1016/S1473-3099(10)70049-9. PMID 20417416
- [Background] Klein SL, Marriott I, Fish EN. Sex-based differences in immune function and responses to vaccination. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):9-15. doi: 10.1093/trstmh/tru167. PMID 25573105
- [Background] Flanagan KL. Vaccines have sex differential non-targeted heterologous effects: a new dawn in vaccine research. Trans R Soc Trop Med Hyg. 2015 Jan;109(1):1-2. doi: 10.1093/trstmh/tru188. No abstract available. PMID 25573102
- [Background] Flanagan KL, van Crevel R, Curtis N, Shann F, Levy O; Optimmunize Network. Heterologous ("nonspecific") and sex-differential effects of vaccines: epidemiology, clinical trials, and emerging immunologic mechanisms. Clin Infect Dis. 2013 Jul;57(2):283-9. doi: 10.1093/cid/cit209. Epub 2013 Apr 9. PMID 23572484
- [Background] Agergaard J, Nante E, Poulstrup G, Nielsen J, Flanagan KL, Ostergaard L, Benn CS, Aaby P. Diphtheria-tetanus-pertussis vaccine administered simultaneously with measles vaccine is associated with increased morbidity and poor growth in girls. A randomised trial from Guinea-Bissau. Vaccine. 2011 Jan 10;29(3):487-500. doi: 10.1016/j.vaccine.2010.10.071. Epub 2010 Nov 18. PMID 21093496

RESULTS

PARTICIPANT FLOW:
Groups:
- MV at 9 Months: All vaccines given as per normal Gambia schedule until 9 months of age, including third dose of diphtheria-tetanus-whole cell pertussis (DTP3), hepatitis B vaccine (HBV) and oral polio vaccine (OPV) at four months of age.
  At 9 months of age given a single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid. Yellow fever vaccine (YF) and OPV administered at 11 months of age. Given a standard MV challenge at 18 months of age.
  Measles Vaccine at 9 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 9 months of age
  Measles Vaccine at 18 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 18 months of age
- DTP + MV at 9 Months: DTP3 dose withheld and given HBV and OPV at four months of age. At 9 months of age given a single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid, and i.m. DTP (Serum Institute of India Ltd.) in the thigh. Yellow fever vaccine (YF) and OPV administered at 11 months of age. Given a standard MV challenge at 18 months old.
  Measles Vaccine at 9 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 9 months of age
  Diphtheria-tetanus-whole cell pertussis vaccine at 9 months of age: Single intramuscular (i.m.) dose of DTP (Serum Institute of India Ltd.) into the thigh at 9 months of age
  Measles Vaccine at 18 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the de
- DTP at 9 Months: DTP3 dose withheld and given HBV and OPV at four months of age. At 9 months of age given i.m. DTP (Serum Institute of India Ltd.) in the thigh. MV, OPV and YF administered at 11 months of age. Given a standard MV challenge at 18 months of age.
  Diphtheria-tetanus-whole cell pertussis vaccine at 9 months of age: Single intramuscular (i.m.) dose of DTP (Serum Institute of India Ltd.) into the thigh at 9 months of age
  Measles Vaccine at 18 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 18 months of age
Period: Overall Study
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Started | 106 | 115 | 81
Completed | 95 | 98 | 68
Not Completed | 11 | 17 | 13
Not completed — Death | 1 | 2 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 2
Not completed — Protocol Violation | 1 | 2 | 3
Not completed — Lost to Follow-up | 3 | 6 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Poor Attendance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- DTP + MV at 9 Months: DTP3 dose withheld and given HBV and OPV at four months of age. At 9 months of age given a single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid, and i.m. DTP (Serum Institute of India Ltd.) in the thigh. Yellow fever vaccine (YF) and OPV administered at 11 months of age. Given a standard MV challenge at 18 old.
  Measles Vaccine at 9 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the deltoid at 9 months of age
  Diphtheria-tetanus-whole cell pertussis vaccine at 9 months of age: Single intramuscular (i.m.) dose of DTP (Serum Institute of India Ltd.) into the thigh at 9 months of age
  Measles Vaccine at 18 months of age: Single standard intramuscular (i.m.) dose of measles vaccine (MV) (Edmonston Zagreb strain, Serum Institute of India Ltd., Pune, India) into the de
- Total: Total of all reporting groups
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months | Total
Number analyzed (Participants) | 106 | 115 | 81 | 302
Age, Continuous [Mean (Standard Deviation); unit: days] | 125 (8) | 124 (7) | 124 (7) | 124 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 56 | 37 | 141
  Male | 58 | 59 | 44 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Group of Mother: Mandinka | 80 | 88 | 56 | 224
  Ethnic Group of Mother: Wolof | 6 | 6 | 5 | 17
  Ethnic Group of Mother: Fula | 9 | 10 | 10 | 29
  Ethnic Group of Mother: Jola | 5 | 3 | 4 | 12
  Ethnic Group of Mother: Other | 6 | 8 | 6 | 20
Region of Enrollment [Number; unit: participants]
  Gambia | 106 | 115 | 81 | 302

OUTCOME MEASURES:

1. Primary Outcome: Effect on Interferon (IFN)-Gamma : Interleukin (IL)-4 Ratio in Plasma
Description: The IFN-gamma:IL-4 cytokine ratio in plasma samples taken 4 weeks after vaccination measured by multiplex assay using the Bio-Plex 200 Suspension Array system. Ratio compared between the 3 intervention groups with the hypothesis that the MV+DTP group will have a higher ratio than the other 2 groups.
Time Frame: 4 weeks after vaccination
Population: Not all participants had this assay done due to the follow reasons: failure to attend the appointment, unwell on the day of follow up, dropped out of the study, assay failure, insufficient blood sample volume or quality.
Measure: Mean (Standard Deviation); unit: ratio of cytokines in pg/mL
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 76 | 78 | 53
ratio of cytokines in pg/mL | 1.48 (1.41) | 1.44 (1.44) | 0.46 (0.58)

2. Primary Outcome: Effect on CD4+FOXP3+CD127- Regulatory T Cell Frequencies
Description: Regulatory T cell (Treg) frequencies (among all gated CD4+ T cells) at 9 and 10 months of age determined by flow cytometry and compared between the 3 intervention groups with the primary hypothesis that the MV+DTP group will have lower Treg frequencies than the MV group.
Time Frame: 4 weeks (9 months and 10 months of age)
Population: Study infants at 9 and 10 months of age. Not all participants had this assay done due to the follow reasons: failure to attend the appointment, unwell on the day of follow up, dropped out of the study, assay failure, insufficient blood sample volume or quality.
Measure: Mean (Standard Deviation); unit: Percentage of CD4+ T cells
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 68 | 77 | 49
Percentage of CD4+ T cells
  9 month values | 5.84 (2.24) | 4.94 (2.24) | 5.86 (1.82)
  10 month values | 6.71 (4.68) | 5.38 (1.87) | 4.85 (2.06)

3. Secondary Outcome: Effect of Vaccine Group on Measles Antibody Levels
Description: Effect of combining MV and DTP on measles antibody responses to see if combining vaccines interferes with antibody generation. Plasma measles antibodies measured by haemagglutination inhibition assay at 9 and 10 months of age.
Time Frame: 4 weeks (9 and 10 months of age)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Haemagglutination titre
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 100 | 110 | 73
Haemagglutination titre
  Value at 9 months of age | 0.29 (0.94) | 0.21 (0.72) | 0.3 (0.96)
  Value at 10 months of age | 5.28 (2.27) | 5.52 (2.18) | 0.37 (1.46)

4. Secondary Outcome: Effect of Vaccine Group on Effector Memory T Cells (TEM)
Description: CD4+CD45RO+CD62L- effector memory T cells measured by flow cytometry at 9 and 10 months of age
Time Frame: 4 weeks (9 and 10 months of age)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent of all CD4+ T cells
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 83 | 91 | 56
Percent of all CD4+ T cells
  TEM at 9 months of age | 3.54 (4.03) | 2.67 (2.42) | 3.10 (2.90)
  TEM at 10 months of age | 4.50 (5.02) | 5.27 (7.91) | 4.52 (6.62)

5. Secondary Outcome: Effect of Vaccine Group on Diphtheria and Tetanus Antibody Levels
Description: Plasma diphtheria and tetanus toxoid antibodies were measured by multiplex microsphere-based fluorescent immunoassay at 9 and 10 months of age.
Time Frame: 4 weeks (9 and 10 months of age)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 100 | 110 | 74
IU/mL
  Tetanus toxoid antibodies at 9 months | 0.62 (0.63) | 0.80 (0.78) | 0.86 (0.90)
  Tetanus antibodies toxoid at 10 months | 0.87 (1.02) | 5.45 (6.24) | 6.46 (5.42)
  Diphtheria toxoid antibodies at 9 months | 0.14 (0.16) | 0.07 (0.10) | 0.13 (0.41)
  Diphtheria toxoid antibodies at 10 months | 0.23 (0.50) | 1.79 (3.02) | 1.57 (1.51)

6. Secondary Outcome: Effect of Vaccine Group on Pertussis Toxoid Antibody Levels
Description: Plasma pertussis toxoid antibodies were measured by multiplex microsphere-based fluorescent immunoassay at 9 and 10 months of age
Time Frame: 4 weeks (9 and 10 months of age)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: EU/mL
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 100 | 110 | 74
EU/mL
  Pertussis toxoid antibodies at 9 months | 18.30 (36.11) | 10.68 (32.15) | 11.11 (37.18)
  Pertussis toxoid antibodies at 10 months | 18.91 (42.31) | 103.72 (149.94) | 86.96 (117.44)

7. Secondary Outcome: Measles Antibody Levels at 19 Months of Age
Description: Measles antibody levels were measured by haemagglutination inhibition assay (HAI) at 19 months of age, 4 weeks after MV challenge at 18 months of age. The aim was to determine whether the vaccination schedule at 9 months of age altered responses to a subsequent MV challenge at 18 months of age i.e., the antibody measurement was made 10 months after the first study intervention.
Time Frame: 10 months (19 months of age)
Population: Study children at 19 months of age. Not all participants had this assay done due to the follow reasons: failure to attend the appointment, unwell on the day of follow up, dropped out of the study, assay failure, insufficient blood sample volume or quality.
Measure: Mean (Standard Deviation); unit: HAI titre
Arm/Group | MV at 9 Months | DTP + MV at 9 Months | DTP at 9 Months
Number analyzed (Participants) | 75 | 78 | 60
HAI titre | 7.74 (1.67) | 7.47 (2.40) | 7.69 (1.25)

ADVERSE EVENTS:
Time Frame: 10 months (from 9 months of age to 19 months of age)
Description: Infants were followed up monthly for 10 months and a clinical questionnaire was completed at each visit.
Groups:
- MV Vaccination at 9 Months: Infants administered MV at 9 months of age
- DTP and MV Vaccination at 9 Months: Infants administered MV and DTP vaccines at 9 months of age
- DTP Vaccination at 9 Months: Infants administered DTP vaccine at 9 months of age
Arm/Group | MV Vaccination at 9 Months | DTP and MV Vaccination at 9 Months | DTP Vaccination at 9 Months
All-Cause Mortality (participants affected / at risk) | 1/106 | 2/115 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/106 | 0/115 | 0/81
Other Adverse Events (participants affected / at risk) | 88/106 | 90/115 | 66/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV Vaccination at 9 Months (N=106) | DTP and MV Vaccination at 9 Months (N=115) | DTP Vaccination at 9 Months (N=81)
Hospital admission with fever and rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV Vaccination at 9 Months (N=106) | DTP and MV Vaccination at 9 Months (N=115) | DTP Vaccination at 9 Months (N=81)
Fever (Infections and infestations) | 19 (25) | 24 (30) | 12 (16) — Fever of unknown cause
Chest infection (Respiratory, thoracic and mediastinal disorders) | 61 (132) | 76 (179) | 48 (99)
Rash, sores (Skin and subcutaneous tissue disorders) | 34 (48) | 36 (49) | 29 (35)
Diarrhoea and / or vomiting (Gastrointestinal disorders) | 56 (97) | 64 (106) | 37 (77)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes